CLINICAL TRIAL: NCT05009485
Title: A Pre-post Intervention Study Evaluating Home-based Management of Patients With Chronic Obstructive Pulmonary Disease or Community Acquired Pneumonia
Brief Title: A Pre-post Intervention Study Evaluating Home-based Management of Patients With COPD or CAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study never started because reprioritization of clinical research efforts
Sponsor: Current Health (Industry)
Collaborators: South Shore Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSH_2021
Record Dates: First submitted 2021-08-10; First posted 2021-08-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Community-acquired Pneumonia
Keywords: wearable; Current Health platform; 30 day readmission
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Community-Acquired Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): Participants will be remotely monitored with the Current Health platform, respond to daily respiratory surveys, receive daily medication reminders and an action plan. Daily dashboard rounds and vital sign alarms from the continuously collected vital signs will be used to identify changes in health and escalated accordingly.
  Interventions: Device: Current Health platform

INTERVENTIONS:
Device: Current Health platform — A remote patient monitoring system which includes a small footprint device and tablet, combined with an AI-powered, cloud-based system driving advanced real-time and predictive analytics related to a patient's clinical condition. The wearable records heart rate, respiratory rate, oxygen saturation, skin temperature and step count.

SUMMARY:
Risk of rehospitalization within 30 days of discharge is higher than 20% in patients with chronic obstructive pulmonary disease (COPD) and up to 20% for patients with community acquired pneumonia (CAP). This pre-post intervention study aims to quantify the impact of continuous remote patient monitoring (RPM) on rates of hospital readmission for patients presenting with CAP or exacerbation of COPD and compare the intervention group to historical controls that did not have access to the intervention. We hypothesize that an intervention combining remote patient monitoring with the remote clinical services and escalation pathways available at SSH (including the Mobile Integrated Health (MIH) program) will reduce hospital readmission within the 30 days following hospital discharge compared to standard of care in this population.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older
* confirmed diagnosis of moderate-severe COPD or community acquired pneumonia
* attendance at South Shore Hospital with an exacerbation of COPD / CAP
* fit for discharge to home

Exclusion Criteria:

* suspicion of COVID-19 or confirmed COVID-19 positive
* life-threatening exacerbation requiring invasive ventilation or prolonged stay in critical care (> 24 hours)
* unable/unwilling to use Current Health
* bilateral axillary lymph node dissection
* persistent atrial fibrillation
* heavy tattooing on upper arms
* discharged to skilled nursing facility
* no access to home or mobile telephone

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a hospital readmission | up to 30 days

SECONDARY OUTCOMES:
Time to service use | up to 30 days
Rate of clinical visits | up to 30 days
  telehealth and/or ambulatory visits
Length of Stay | up to 30 days
  original and subsequent readmissions or emergency department attendance
Rate of Mortality | up to 30 days
Rate of medication adherence | up to 30 days
Progression of Disease | up to 30 days
  medication requirements, oxygen dependence, spirometric changes

OTHER OUTCOMES:
Patient Satisfaction as assessed by the Telehealth Usability Questionnaire | up to 30 days
  subdomain of the Telehealth Usability Questionnaire that includes 4 questions measured on a 7-point Likert scale.

IPD SHARING:
Plan to Share IPD: Undecided